CLINICAL TRIAL: NCT03266003
Title: An Evaluation of Traditional Directly Observed Therapy and Electronic Forms of Directly Observed Therapy for Tuberculosis Treatment
Brief Title: An Evaluation of Traditional Directly Observed Therapy (DOT) and Electronic DOT for TB Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: New York City Department of Health and Mental Hygiene (Other Government); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: CDC-6995.0
Record Dates: First submitted 2017-07-26; First posted 2017-08-29 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Tuberculosis; Drug-resistant Tuberculosis; Adherence, Medication; Adherence, Patient
Keywords: Tuberculosis; Directly observed therapy; Adherence; Video assisted directly observed therapy; Electronic directly observed therapy; Mobile health
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant; Medication Adherence; Patient Compliance; Directly Observed Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: ipDOT followed by eDOT (Other): Following 20 observable medication doses under an initial DOT study group assignment of in-person DOT (ipDOT), patients will be assigned (crossed-over) to electronic DOT (eDOT) to collect data on another 20 observable medication doses.
  Interventions: Other: Electronic DOT; Other: In-person DOT
- Group 2: eDOT followed by ipDOT (Other): Following 20 observable medication doses under an initial DOT study group assignment of electronic DOT (eDOT), patients will be assigned (crossed-over) to in-person DOT (ipDOT) to collect data on another 20 observable medication doses.
  Interventions: Other: Electronic DOT; Other: In-person DOT

INTERVENTIONS:
Other: Electronic DOT — Electronic DOT is the use of electronic communication methods to observe patients swallow anti-TB drugs and monitor for medication side effects. This study will use two variations of electronic communication methods, referred to as "electronic directly observed therapy" or "eDOT". This includes: (1) eDOT conducted "live" in which TB program staff interact with patients via a computer or phone application as they ingest their medication (eDOT-live), and (2) eDOT conducted using "time stamped, recorded" videos in which TB program staff log into an electronic system and review videos recorded by patients in order to verify that patients ingested their medication doses as scheduled (eDOT-recorded).
  Other Names: eDOT; Video DOT (VDOT)
Other: In-person DOT — A trained person is in the physical presence of patients as anti-TB drugs are ingested.
  Other Names: ipDOT; Traditional DOT

SUMMARY:
This study is a U.S.-based, 1 site (with 4 clinical settings), randomized controlled trial (with funding from the Centers for Disease Control and Prevention's (CDC) Antibiotic Resistance Solutions Initiative) that will be implemented to evaluate traditional directly observed therapy (DOT) and electronic forms of DOT (eDOT) for tuberculosis (TB) treatment. The trial will assess whether eDOT that employs electronic communication methods, such as video via computer or cellphone, is a non-inferior approach to monitor TB treatment adherence, compared to traditional in-person DOT (ipDOT), in which a trained person is in the physical presence of patients as anti-TB drugs are ingested. ipDOT is the single best intervention proven to be successful when it comes to TB patients' adherence to therapy (which reduces risk of acquired drug resistance). However, ipDOT is resource intensive and many times challenging to facilitate in-person. If eDOT is found to be non-inferior to ipDOT, health departments and other clinicians might be able to provide eDOT to certain populations of TB patients in a more flexible and potentially cost-saving manner.

DETAILED DESCRIPTION:
Tuberculosis (TB) is among the most common infectious diseases and cause of death worldwide. The bacteria that causes TB, Mycobacterium tuberculosis (Mtb), is spread when a person with TB disease of the lungs or throat coughs, speaks, or sings. These bacteria can float in the air for several hours, depending on the environment. Persons who breathe in the air containing these TB bacteria can become infected.

The World Health Organization (WHO) estimates that 9.6 million became ill with TB in 2014. Among this group, approximately 480,000 persons became ill with multidrug-resistant TB (MDR TB), which is TB caused by bacteria that are resistant to at least isoniazid and rifampin, the two most potent TB drugs used to treat persons with TB disease. Extensively drug resistant (XDR) strains of TB were reported by 105 countries in 2015. As such, the National Strategy for Combatting Antibiotic Resistant Bacteria (CARB) has designated Mtb a SERIOUS threat level pathogen.

Completion of treatment by persons with TB disease represents the optimal path to the prevention of morbidity and mortality, cure of the patient, interruption of transmission, and prevention of acquired drug resistance. The single best intervention in this regard has proven to be directly observed therapy (DOT).

DOT provides frequent interactions between the patient and the patient's healthcare team. This enables better monitoring and efficient response to medication side effects. This is especially important as medication side effects are among the top reasons patients are lost to follow-up during treatment therapy.

Experience in the U.S. in the 1990s demonstrated the efficacy of this intervention in the prevention and control of drug-resistant tuberculosis.Studies in the past 15 years in international settings have challenged the utility of DOT, but have been criticized for imperfect to poor design or implementation.

DOT entails a trained "observer" acceptable to both the patient and the health system being present to monitor treatment adherence as patients swallow anti-TB drugs. In the United States, DOT remains a cornerstone of TB control. While DOT represents the treatment standard, the implementation of DOT has been modified by some programs in an effort to reduce costs and conserve program resources. In the U.S., efforts recently have sought to utilize advances in communication technology to facilitate the implementation of DOT.

This study will evaluate traditional approaches to DOT compared to DOT by electronic methods. The study will be based within, and primarily conducted by the New York City Department of Health and Mental Hygiene (NYC DOHMH), Bureau of Tuberculosis Control (BTBC) clinics. This will enable the study to be to be conducted in a programmatic setting and reflect "real-life" situations.

Hypothesis: Directly observed therapy (DOT) that employs electronic communication methods (eDOT) is a non-inferior approach to monitor treatment adherence, compared to traditional forms of DOT, in which a trained person is in the physical presence of patients as anti-TB drugs are ingested (ipDOT).

Design: This will be a U.S.-based, 1 site (with 4 clinic settings), randomized, cross-over, 2-arm, non-inferiority trial with randomization to either traditional in-person DOT (ipDOT) or electronic DOT (eDOT)*, at the time outpatient treatment begins within participating health department clinics.

*Secondary analyses will evaluate DOT conducted in "real time" or "live" (eDOT-live) compared to DOT that uses a recorded video (eDOT-recorded).

Population:Patients newly diagnosed with drug-sensitive or non-rifamycin resistant TB.

Site: Four clinics of the New York City Department of Health and Mental Hygiene, Bureau of Tuberculosis Control.

Study Duration: Duration per participant is approximately 6 months.

Description of Intervention: After providing written informed consent, participants will be randomly assigned to one of the following DOT study group assignments: (1) traditional in-person DOT (ipDOT) or (2) electronic DOT (eDOT).

Note: Patients and their providers will discuss and choose the type of eDOT they will use. The two options are: (2a) eDOT conducted "live" in which TB program staff interact with patients in real-time via a computer or phone application as they ingest their medication (eDOT-live), and (2b) eDOT in which patients record themselves ingesting their TB medication using "time-stamped, recorded" videos for TB program staff to review within 1 business day (24 hours), and verify that patients ingested their medication doses as scheduled (eDOT-recorded).

Following 20 observable medication doses under an initial DOT study group assignment participants will be assigned (crossed-over) to the opposite DOT method to collect data on another 20 observable medication doses. Specifically, participants who initially received ipDOT will switch to eDOT. Participants initially assigned to eDOT will switch to ipDOT.

At the conclusion of this Cross-Over Period with 40 observable medication doses, participants will continue treatment using their preferred DOT method.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet the following inclusion criteria in order to participate in this study:

1. All TB patients (both those with a confirmed diagnosis and those with a clinical diagnosis), started on treatment for non-rifamycin resistant TB, and eligible to receive DOT.
2. Physician determines the patient may be treated with any treatment regimen for non-rifamycin resistant TB approved by the NYC DOHMH TB program.
3. Individuals found to have Isoniazid (INH) resistant disease are eligible for inclusion.
4. Age >18 years or older
5. Age 12 to 17 years, with the consent of a parent or legal guardian
6. An address or residence location that is readily accessible for visiting, and willingness to inform the study team of any change of address during the treatment and follow-up period.
7. No plans to move out of the catchment areas of the participating TB program sites within 9 months of enrollment.
8. Willingness to comply with study procedures and provide written informed consent prior to study enrollment.
9. Individuals for whom a diagnosis of TB has been made clinically are eligible for study inclusion. Data may be collected from these patients related to all objectives with the exception of culture conversion.

Exclusion Criteria:

An individual meeting any of the following exclusion criteria at the time of enrollment will be excluded from study participation:

1. At the time of enrollment, the patient's Mtb isolate is already known to be resistant to rifamycin or prescribed a non-rifamycin treatment regimen.
2. Prescribed any injectable, anti-TB medication as part of an outpatient treatment regimen.
3. Adverse reaction to initial doses of anti-TB medication (per NYC protocol) of sufficient severity that in the judgement of the clinician makes study participation not in the individual's best interest.
4. A cognitive or physical disability that prevents full participation in eDOT (e.g., vision, hearing, physically challenged, inability to swallow medications). Note: Exceptions will be made for those patients who crush pills in order to swallow the medication, or have a member of their household or a caregiver who can assist them for the duration of the study.
5. Less than 12 years of age.
6. Patients 12-17 years of age, whose parents or legal guardians refuse to provide consent.
7. Incarceration, institutionalization, or other involuntary detention.
8. Plans to move out of the catchment areas of the participating TB program sites in less than 9 months from the day of enrollment.
9. Previously enrolled in this study.
10. Currently enrolled in a clinical trial that prohibits enrollment in another study.
11. Other medical conditions that, in the investigator's or the clinic physician's judgment, make study participation not in the individual's best interest.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of medication doses directly observed | 6 months
  The proportion of medication doses that are directly observed by staff.

SECONDARY OUTCOMES:
Proportion of medication doses not directly observed | 6 months
  The proportion of medication doses not directly observed due to equipment malfunction or loss, staff unavailability, patient travel/ work/ school, inclement weather, or other reasons.
Medication side effects | Up to 13 weeks
  Time, measured in days, in which participants experience initial symptoms of medication side effects to when they receive medical attention for the medication side effects they are experiencing, either through consultation with a physician, urgent care or emergency room visits, or hospital admission across DOT methods.

OTHER OUTCOMES:
Patients' demographic, social, and medical characteristics associated with treatment adherence | 6 months
  Number of participants by gender, race, ethnic origin, country of birth, primary language spoken, and employment who adhere to TB treatment. Additionally, the number of patients with a history of contact with persons diagnosed with multi-drug resistant TB, incomplete treatment for latent TB infection, diabetes, renal disease, immunosuppression, hepatitis, a history of homelessness, a history of substance abuse, a history of incarceration, a history of a prior TB diagnosis who adhere to TB treatment.
Treatment outcomes | 6 months
  Compare the proportion of participants completing treatment to those lost to follow-up or refused further treatment, transfer or move, experience treatment failure, or expire (with death attributable to tuberculosis) across DOT methods.
Participants' preferred DOT method at the conclusion of the cross-over period. | 8 -13 weeks
  After participants complete 40 doses of TB medication (20 doses using ipDOT and 20 doses using eDOT) during the cross-over period, they will be asked to report which DOT method they prefer, and the reasons for their preference.
Patient Opinion Questionnaire | 8-13 weeks
  After participants complete 40 doses of TB medication (20 doses using ipDOT and 20 doses using eDOT), participants will be asked to complete the Patient Opinion Questionnaire to assess their perceptions of the quality of care across DOT methods and satisfaction with patient-staff relationships/rapport.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Burzynski, MD, MPH, Principal Investigator — New York City DOHMH, Bureau of Tuberculosis Control
Locations (4):
- United States (4):
  - Fort Greene Chest Center, Brooklyn, New York
  - Corona Chest Center, Jackson Heights, New York
  - Washington Heights Chest Center, New York, New York
  - Morrisania Chest Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: Undecided
Any proposal for additional analysis of study data must be agreed to in advance by the NYC DOHMH BTBC and CDC investigators.
  These criteria will not apply to public-use data that have been made available in accordance with CDC's policy on data sharing. Persons who use publicly available data will be asked to acknowledge both the NYC DOHMH BTBC and CDC.

REFERENCES:
- [Derived] Mangan JM, Burzynski J, deCastro BR, Salerno MM, Lam CK, Macaraig M, Reaves M, Kiskadden-Bechtel S, Bowers S, Sathi C, Dias MP, Goswami ND, Vernon A. Challenges associated with electronic and in-person directly observed therapy during a randomized trial. Int J Tuberc Lung Dis. 2023 Apr 1;27(4):298-307. doi: 10.5588/ijtld.22.0583. PMID 37035970
- [Derived] Burzynski J, Mangan JM, Lam CK, Macaraig M, Salerno MM, deCastro BR, Goswami ND, Lin CY, Schluger NW, Vernon A; eDOT Study Team. In-Person vs Electronic Directly Observed Therapy for Tuberculosis Treatment Adherence: A Randomized Noninferiority Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2144210. doi: 10.1001/jamanetworkopen.2021.44210. PMID 35050357